CLINICAL TRIAL: NCT05793905
Title: Evaluation of the Effect of Buffered Anesthetic Solution (Lidocaine 2%) in the Effectiveness of Inferior Alveolar Nerve Block Injection During the Treatment of Mandibular Primary Molars
Brief Title: Buffered Anesthetic Solution in the Treatment of Mandibular Primary Molars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UDDS-Pedo-03-2023
Record Dates: First submitted 2023-02-07; First posted 2023-03-31 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Local Anesthesia
Keywords: Buffered lidocaine
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: This clinical research aims to evaluate the effectiveness of buffered lidocaine in the treatment of bilateral primary molars
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple Masking: Patients, Investigators and Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buffered lidocaine (Experimental): Inferior alveolar nerve block with buffered anesthetic solution (2% lidocaine with 1/80000 adrenaline mixed with sodium bicarbonate 8.4%)
  Interventions: Combination Product: Buffered lidocaine in inferior alveolar nerve block injection
- Lidocaine 2% (Other): Control group:
  Inferior alveolar nerve block with anesthetic solution (Lidocaine 2% with adrenaline 1.80000).
  Interventions: Drug: lidocaine 2% in inferior alveolar nerve block injection

INTERVENTIONS:
Combination Product: Buffered lidocaine in inferior alveolar nerve block injection — Buffered Lidocaine 2% with epinephrine 1.80000 mixed with 1.8% sodium bicarbonate in IANB injection in the treatment of bilateral primary mandibular molars
  Other Names: Buffered lidocaine
  Arms: Buffered lidocaine
Drug: lidocaine 2% in inferior alveolar nerve block injection — Lidocaine 2% with epinephrine 1.80000 in IANB injection in the treatment of bilateral primary mandibular molars
  Arms: Lidocaine 2%

SUMMARY:
In a prospective, randomized clinical trial, triple-blind, split-mouth study, 40 children aged between 7 to 10 with bilateral mandibular primary molars were diagnosed with pulpitis. The test agent was 2% lidocaine with 1:80.000 epinephrine buffered with sodium bicarbonate 8.4% at a ratio of 1/10, as opposed to the control agent, which was non- buffered 2% lidocaine with 1:80,000 epinephrine. The pain will be assessed during inferior alveolar nerve block injection (IANB) and the effectiveness of anesthesia using the subjective Wong-Baker visual analog scale, the objective sound, eye, and motor (SEM) scale, and the physiological pain scale (pulse rate) using a pulse oximeter. The investigator has confirmed the onset of anesthesia after lip tongue-numbing by probing the gingiva until there is no pain. Endo-ice has been used to assess the onset of pulp anesthesia.

DETAILED DESCRIPTION:
In a prospective, randomized clinical trial and triple-blind, split mouth study, 40 children aged between 7 to 10 with bilateral mandibular primary molars were diagnosed with pulpitis. Random numbers between 1 to 40 were assigned to patients, with some receiving buffered lidocaine at their initial appointment while others received unbuffered lidocaine. The solutions have been switched up for the second session, which has been set for one week later. The test agent was 2% lidocaine with 1:80.000 epinephrine buffered with sodium bicarbonate 8.4% at a ratio of 1/10, as opposed to the control agent, non-buffering 2% lidocaine with 1:80,000 epinephrine. Buffered lidocaine has been freshly prepared by mixing sodium bicarbonate (8.4%) with the anaesthetic solution (lidocaine 2% with epinephrine 1/80.000) in a 1:10 ratio by volume. Two percent benzocaine gel is applied at the injection site for one minute before inferior alveolar nerve block injection (IANB). The investigator has assessed pain during IANB injection using the subjective Wong-Baker visual analogue scale, the objective sound, eye, and motor (SEM) scale, and the physiological pain scale (pulse rate) using a pulse oximeter. After administering the IANB injection, the investigator has confirmed the onset of anaesthesia after lip and tongue numbing by probing the gingiva every 30 seconds until there is no pain. Endo-ice has been used to assess the onset of pulp anaesthesia every 30 seconds. The effectiveness of anaesthesia has been assessed during the preparation of the pulp chamber using subjective, objective, and physiological pain scales. Finally, the numerical data will be statistically analysed, and any statistically significant values will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Children who are healthy and free of any underlying conditions that might make local anesthesia impossible to administer.
* Children that are not allergic to (lidocaine, adrenaline, or sodium bicarbonate).
* Children aged 6-10 years old
* Cooperative children on Frankel scale (positive or absolute positive).
* children needing bilateral (right and left) endodontic treatment for the mandibular primary molars.
* A positive outcome on the cold test for the target tooth.

Exclusion Criteria:

* Uncooperative children on Frankel's scale (passive or absolute positive).
* The presence of a fistula.
* The presence of an abscess associated with the target tooth.
* The presence of a periapical lesion radially.
* Negative response to the cold test.
* Children suffering from systemic conditions.
* Children who are allergic to (lidocaine, adrenaline, sodium bicarbonate).

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Probing the gingiva | directly after asking the child about lip, tongue numbing every 30 seconds until there is no pain.
  The onset of anaesthesia at soft tissue will be assessed by probing the gingiva After IANB injection.
Endo - ice test | Every 30 seconds after confirmed soft tissues anaesthesia until the absence of pain.
  The investigator will use endo-ice to assess the onset time of pulp anaesthesia.
Pulse rate | A minute before anaesthesia.
  Pulse rate is a physiological pain scale which will be taken through a finger pulse oximeter.
Pulse rate | 20 seconds after the first quarter of the local anaesthesia.
  Pulse rate is a physiological pain scale, will be taken through a finger pulse oximeter.
Wong baker faces scale. | One minute after IANB injection
  Wong Baker faces scale is a subjective pain which contains a series of six faces ranging from a happy face at 0 to indicate "no hurt" to a crying face at 10 to indicate "hurts worst"
Sound, eye, motor scale (SEM) | Within five seconds from the start of the local anesthetic injection to completion
  Sound, eye, motor scale is an objective pain scale for the assessment of child's behaviour by recording video during anaesthesia

SECONDARY OUTCOMES:
Pulse rate | 20 seconds after opening the pulp chamber
  Pulse rate is a physiological pain scale which will be taken through a finger pulse oximeter.
Wong baker faces scale | one minute after preparing pulp chamber
  Wong Baker faces scale is a subjective pain which contains a series of six faces ranging from a happy face at 0 to indicate "no hurt" to a crying face at 10 to indicate "hurts worst"
sound, eye, motor scale (SEM) | Within five seconds from the start of the local anaesthetic injection to completion
  Sound, eye, motor scale is an objective pain scale for the assessment of child's behaviour by recording video during endo access preparation

CONTACTS AND LOCATIONS:
Overall Officials: Chaza Kouchaji, Professor, Study Director — Supervisal; Hanadi Almattit, Phd,lecturer, Study Director — Co- supervisal
Locations (1):
- College of dentistry., Damascus, Al-Mazzeh Saint, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chopra R, Jindal G, Sachdev V, Sandhu M. Double-Blind Crossover Study to Compare Pain Experience During Inferior Alveolar Nerve Block Administration Using Buffered Two Percent Lidocaine in Children. Pediatr Dent. 2016 Jan-Feb;38(1):25-9. PMID 26892211
- [Result] Goodchild JH, Donaldson M. Novel Direct Injection Chairside Buffering Technique for Local Anesthetic Use in Dentistry. Compend Contin Educ Dent. 2019 Jul/Aug;40(7):e1-e10. PMID 31478693
- [Result] Meincken M, Norman C, Arevalo O, Saman DM, Bejarano T. Anesthesia Onset Time and Injection Pain Between Buffered and Unbuffered Lidocaine Used as Local Anesthetic for Dental Care in Children. Pediatr Dent. 2019 Sep 15;41(5):354-357. PMID 31648665
- [Result] Kurien RS, Goswami M, Singh S. Comparative evaluation of anesthetic efficacy of warm, buffered and conventional 2% lignocaine for the success of inferior alveolar nerve block (IANB) in mandibular primary molars: A randomized controlled clinical trial. J Dent Res Dent Clin Dent Prospects. 2018 Spring;12(2):102-109. doi: 10.15171/joddd.2018.016. Epub 2018 Jun 20. PMID 30087760